CLINICAL TRIAL: NCT05869500
Title: Left Bundle Area Pacing Vs. Right Ventricular Pacing in Patients With Normal Left Ventricular Function -The Boston Pace Study
Brief Title: The Boston Pace Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Chee Yuan Ng, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022P003143
Record Dates: First submitted 2023-04-17; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Left Bundle Branch Area Pacing
Keywords: left bundle branch; left bundle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Left Bundle Branch Area Pacing (Experimental)
  Interventions: Device: Left Bundle Branch Area Pacemaker
- Right Ventricular Pacing (Active Comparator)
  Interventions: Device: Right Ventricular Pacemaker

INTERVENTIONS:
Device: Left Bundle Branch Area Pacemaker — Implantation of Medtronic 3830 lead for left bundle branch area pacing
  Arms: Left Bundle Branch Area Pacing
Device: Right Ventricular Pacemaker — Implantation of a conventional right ventricular pacemaker lead
  Arms: Right Ventricular Pacing

SUMMARY:
Right ventricular (RV) pacing can cause left ventricular systolic dysfunction in 10- 20% of patients. Biventricular pacing had previously been shown to prevent left ventricular systolic dysfunction. However, implantation of coronary sinus lead increases procedural risk and can be limited by higher threshold and phrenic nerve capture. HIS pacing has been evaluated as an alternative pacing strategy, but its routine use was limited by difficulty of the procedure, success rate and high pacing threshold.

Left bundle branch area pacing (LBBAP) is a promising physiologic pacing technique that has been proposed as a pacing strategy to prevent pacing induced cardiomyopathy and for treatment of desynchrony in heart failure. LBBAP has been adopted widely and performed routinely on patients with AV block. Currently, it is up to the discretion of the proceduralist whether LBBAP is performed given that there is lack of evidence to guide pacing strategies.

DETAILED DESCRIPTION:
This pilot trial is a feasibility study that will assess for efficacy, safety and success rate of left bundle branch area pacing. The study will also examine the recruitment rate at 2 major tertiary hospitals.

The study will examine if the use of LBBAP can prevent the occurrence of pacing induced cardiomyopathy (PICM) compared to RV pacing among patients with normal left ventricular function and high-grade AV block.

The investigators hypothesize that the rate of pacing induced cardiomyopathy is lower with LBBAP compared to RV pacing in patients with normal left ventricular function requiring high burden of RV pacing.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Patients with complete AV block, high-grade AV block with an anticipated ventricular pacing rate of more than 40%
3. Left ventricular ejection fraction of 50% or more.
4. Echocardiogram within the last 3 months

Exclusion Criteria:

1. History of systolic dysfunction with LV EF of less than 50%
2. Prior myocardial infarction
3. Obstructive coronary artery disease
4. Severe valvular dysfunction
5. Life expectancy of less than a year
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF) | 12 months
Change in left ventricular end systolic volume (LVESV) | 12 months

SECONDARY OUTCOMES:
Success rate of LBBAP | 30 days
All-cause mortality | 12 months
Cardiovascular mortality | 12 months
Rate of heart failure related visit: defined as heart failure hospitalization or emergency room visit or urgent visit requiring intravenous heart failure therapy | 12 months
Number of participants with upgrade to cardiac resynchronization therapy | 12 months
New York Heart Association Class I-IV (IV is worst) | 12 months
Number of participants with occurrence of moderate or severe tricuspid regurgitation on echocardiogram | 12 months
Number of participants with occurrence of moderate or severe mitral regurgitation on echocardiogram | 12 months
Number of participants with new onset atrial fibrillation | 12 months
Kansas City Cardiomyopathy Questionnaire (KCCQ-12) (score of 8-40) | 12 months
Paced QRS duration on 12 lead EKG | Evaluated at 1 day, 30 days and 12 months
Pacing percentage | 12 months
Complication rate including pneumothorax, cardiac tamponade, infection, and lead revision | 12 months
Procedure time | 1 day
Fluoroscopy time | 1 day
Pacing capture threshold (V) | 12 months
R wave amplitude (mV) | 12 months
RV lead impedance (ohms) | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided